CLINICAL TRIAL: NCT02177188
Title: HEAVy HAT-HEAlthy Volunteers Heart to Arm Time. Haemorrhage Simulation Protocol in Healthy Volunteers.
Acronym: HEAvyHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HHAT2012
Record Dates: First submitted 2013-03-01; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Shock
Keywords: Hypovolaemic shock; Monitoring; Haemorrhage; Transthoracic Echocardiography
MeSH Terms: conditions — Shock; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haemorrhage simulation (Experimental)
  Interventions: Device: LBNP Lower Bodi Negative Pressure Chamber

INTERVENTIONS:
Device: LBNP Lower Bodi Negative Pressure Chamber

SUMMARY:
In prehospital settings, hypovolemic shock diagnosis is based on Advanced Trauma Life Support (ATLS) shock classification. The most often used clinical signs are heart rate (HR), arterial blood pressure (BP), respiratory rate, neurologic status, diuresis, skin colour and temperature. However, some of these signs, such as hypotension and tachycardia, lack specificity and sensitivity and do not occur early enough. Even with an early preload reduction, blood pressure can remain constant due to compensatory mechanisms, such as vasoconstriction and positive chronotropism. Tachycardia occurs earlier, but has poor specificity and sensitivity. A retrospective analysis of 25,287 trauma patients showed that among 489 patients presenting with systolic BP < 90 mmHg, only 65% had tachycardia (HR > 90 bpm), while 39% of patients with systolic BP > 120 mmHg were tachycardic, probably resulting from other stimuli influencing heart rate, such as pain, fear, circulating hormones and endogenous enkephalins. Therefore, it could be very useful to have an index that identifies initial volume variation, when physiological regulatory mechanisms are still effectively maintaining normal BP.

Pulse transit time (PTT) is the sum of pre-ejection period (PEP; the time interval between the onset of ventricular depolarization and ventricular ejection) and vascular transit time (VTT; the time it takes for the pulse wave to travel from the aortic valve to peripheral arteries). PEP and VTT variations depend on preload variation, and PTT increases with PEP, showing a linear correlation (R2 = 0.96). Chan et al. subjected 11 healthy volunteers to the head-up tilt test, and demonstrated that PEP increased and VTT decreased for increasing tilt angles from 0° to 80°, corresponding to light-moderate bleeding. They also observed early sympathetic activation, expressed by decreases of both RR interval (RR) and VTT, dampening the PTT increase, since PTT is influenced by both continuous PEP increase and progressive VTT decrease occurring during hypovolaemia.

Here the investigators describe a new index, called indexed Heart to Arm Time (iHAT). iHAT is the mPTT/RR ratio, where mPTT is a modified PTT, measured from the onset of ventricular depolarization (the 'R' wave of the ECG trace) to the systolic peak of the photoplethysmographic pulse oxymetry (PPG) waveform. mPTT is indexed to RR interval on ECG to counteract sympathetic activation that would dampen PEP increase and enhance VTT reduction, by means of positive inotropism and peripheral vasoconstriction, respectively. iHAT therefore increases during haemorrhage because of preload reduction and the consequent PEP increase and RR interval decrease. iHAT is expressed as the time percentage of the interbeat interval (RR) it takes to the PPG waveform to travel to peripheral arteries. In this study iHAT has been calculated as the average of beat-to-beat mPTT/RR ratios over 30 heart beats (corresponding to at least 2 breathing cycles) in order to minimize the effect of spontaneous breathing on preload, and thus on PEP and PTT.

In the present study, the investigators aimed to evaluate iHAT in a simulating model of hypovolaemia by using a Lower Body Negative Pressure (LBNP) chamber. LBNP chamber simulates haemorrhage by applying negative pressure to the lower limbs, thus giving an accurate model of hypovolemia. The LBNP chamber has been used for many years for research purposes, and in 2001 Convertino suggested it is a useful device to test severe haemorrhage-related hemodynamic responses. In fact, the induced volemic sequestration is an efficient technique to study physiological behaviours in humans.

The primary endpoint was to evaluate the use of the iHAT as a predictor of hypovolaemia. The secondary endpoint was to compare the specificity and sensitivity of the iHAT index compared to commonly used indexes (BP, HR). Furthermore, the investigators aimed to assess feasibility of Transthoracic echocardiography (TTE) evaluation of Cardiac Output (CO) in a haemorrhagic model and to evaluate CO changes with respect to measured hemodynamic variables.

TTE evaluation of CO is non invasive and comparable to thermodilution, and of possible use in an emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* 30 healthy volunteers with no assumption of coffee or any other substance with possible action on the autonomic nervous system.

Exclusion Criteria:

* age < 18 yrs,
* pregnancy,
* assumption of any drugs and existence of any disease,
* intake of any drug/substance with action on the autonomic nervous system during the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
iHAT validation as a bleeding predictor in a simulated and controlled haemorrhage model (Lower Body Negative Pressure chamber, LBNP) | Progressive lower body negative pressure (LBNP) was applied in 5-min stages until the onset of impending cardiovascular collapse.

SECONDARY OUTCOMES:
Change from baseline in CO evaluated by Transthoracic echocardiography (TTE) during an haemorrhagic model | Progressive lower body negative pressure (LBNP) was applied in 5-min stages until the onset of impending cardiovascular collapse.

CONTACTS AND LOCATIONS:
Locations (1):
- AO Ospedale Niguarda Ca' Granda, Milan, Italy

REFERENCES:
- [Background] Chan GS, Middleton PM, Celler BG, Wang L, Lovell NH. Change in pulse transit time and pre-ejection period during head-up tilt-induced progressive central hypovolaemia. J Clin Monit Comput. 2007 Oct;21(5):283-93. doi: 10.1007/s10877-007-9086-8. Epub 2007 Aug 16. PMID 17701385
- [Background] Esch BT, Scott JM, Warburton DE. Construction of a lower body negative pressure chamber. Adv Physiol Educ. 2007 Mar;31(1):76-81. doi: 10.1152/advan.00009.2006. PMID 17327587
- [Background] Convertino VA. Lower body negative pressure as a tool for research in aerospace physiology and military medicine. J Gravit Physiol. 2001 Dec;8(2):1-14. PMID 12365445